CLINICAL TRIAL: NCT03574545
Title: A Randomized, Open Label, Multiple Dose, Parallel Group Study to Assess the Safety and Pharmacokinetic Comparability of Two VAY736 Drug Products in Patients With Rheumatoid Arthritis
Brief Title: Study Comparing Two VAY736 Drug Products in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVAY736A2101; 2018-001173-24 (EudraCT Number)
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; VAY736; Ianalumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ianalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference VAY736 Drug Product (Active Comparator): Powder for solution for injection / infusion
  Interventions: Biological: ianalumab
- Test VAY736 Drug Product (Experimental): Solution for injection
  Interventions: Biological: ianalumab

INTERVENTIONS:
Biological: ianalumab — Human monoclonal antibody (mAb) of type IgG1/κ binding to B-cell activating-receptor (BAFF-R)
  Other Names: VAY736

SUMMARY:
This study will assess the safety and pharmacokinetic comparability of two VAY736 drug products in patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill 2010 ACR/EULAR criteria for RA Aletaha et al 2010 at Screening
* Active disease defined as ≥ 2 swollen joints (of 58 evaluable joints) and ≥ 2 tender joints (of 60 evaluable joints) despite stable MTX ≤ 25 mg/week and/or hydroxychloroquine ≤ 400 mg/day treatment for at least 2 months prior to randomization

Exclusion Criteria:

* Prior or previous use of (specific dosages and intervals prior to study start may apply): other investigational drugs, B-cell depleting therapy (e.g. rituximab), monoclonal antibodies (mAb), i.v. / s.c. Ig, thymoglobulin, i.v. or oral cyclophosphamide, oral cyclosporine, soluble cytokine receptors, azathioprine.
* Currently receiving prednisone >10 mg/day (or equivalent oral glucocorticoid) or dose adjustment within 2 weeks prior to randomization
* Active viral, bacterial or other infections requiring systemic treatment at the time of screening or enrollment, or history of recurrent clinically significant infection or of bacterial infections with encapsulated organisms
* Receipt of live/attenuated vaccine within a 2-month period before randomization
* Pregnant or nursing (lactating) women
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception from screening and for 4 months after stopping of investigational drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by the number of patients with adverse events | Week 0 - 112
  The number of patients with adverse events after repeated subcutaneous (s.c) injections of a fixed dose of ianalumab
Pharmacokinetic comparability at steady state - AUCtau | Week 8 - 12
  The area under the serum ianalumab concentration-time curve from time zero to the end of the dosing interval (AUCtau)
Pharmacokinetic comparability at steady state - Cmax | Week 8 - 12
  Observed maximum serum concentration of ianalumab following drug administration (Cmax)

SECONDARY OUTCOMES:
Pharmacokinetic comparability after the first dose - AUCtau | Week 0 - 4
  The area under the serum ianalumab concentration-time curve from time zero to the end of the dosing interval (AUCtau)
Pharmacokinetic comparability after the first dose - Cmax | Week 0 - 4
  Observed maximum serum concentration of ianalumab following drug administration (Cmax)
Pharmacokinetic comparability after the first dose - Tmax | Week 0 - 4
  Time to reach the maximum concentration after drug administration (Tmax)
Pharmacokinetic comparability of two ianalumab drug products after the last dose - AUCinf | Week 8 - 12
  The area under the serum ianalumab concentration-time curve from time zero to infinity (AUCinf)
Pharmacokinetic comparability after the last dose - Tmax | Week 8 - 12
  Time to reach the maximum concentration after drug administration (Tmax)
Pharmacokinetic comparability after the last dose - T1/2 | Week 8 - 12
  The terminal elimination half-life (T1/2)
Pharmacokinetic comparability at the end of each dosing interval - Ctrough | Week 0 - 12
  Observed minimum serum ianalumab concentration following drug administration (Ctrough)
Pharmacodynamic effect as measured by B-cell level | Week 0 - 112
  Circulating B cells (CD19+)
Immunogenicity as measured by Anti-Drug Antibodies | Week 0 - 112
  Anti-ianalumab antibodies (ADA); incidence of ADA positive patients and correlation with AEs, PK and clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, Berlin, Germany
- Novartis Investigative Site, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to results from the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18328
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2687